CLINICAL TRIAL: NCT02049255
Title: Comparision of the Use in Marcaine and Chloroprocaine in Rachianesthesia for the Surgical Correction of Inguinal Hernia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric DEFLANDRE, MD, FCCP, Astes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMBES-ASTES-2013
Record Dates: First submitted 2014-01-24; First posted 2014-01-30 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: All
MeSH Terms: conditions — Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — chloroprocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marcaine (Placebo Comparator): Rachianesthesia with marcaine or chloroprocaine
  Interventions: Drug: Marcaine
- Chloroprocaine (Active Comparator): Rachianesthesia with marcaine or chloroprocaine
  Interventions: Drug: Chloroprocaine

INTERVENTIONS:
Drug: Chloroprocaine — The Group "Chloroprocaine" will receive: Chloroprocaine: 50 mg in rachianesthesia
  Arms: Chloroprocaine
Drug: Marcaine — The Group "Marcaine" will receive: Marcaine: 12,5 mg in rachianesthesia
  Arms: Marcaine

SUMMARY:
Comparison the use of marcaine and chloroprocaine in rachianesthesia for a surgical correction of inguinal hernia. Comparision between acute and chronic (3 months and 6 months) pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults under rachianesthesia

Exclusion Criteria:

* Personal history of gastric ulcus
* ASA 4
* Emergency
* Combined surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Acute pain | 1 day of the surgery when patient leave the recovery room

SECONDARY OUTCOMES:
Chronic pain | at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Deflandre, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc Bouge, Bouge, Namur, Belgium